CLINICAL TRIAL: NCT01121952
Title: The Effect of Manipulation on Dysfunction of the Talo-crural Joint- a Clinical Randomised Trial
Brief Title: The Effect of Manipulation on Dysfunction of the Talo-crural Joint
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scandinavian College of Chiropractic (Other)
Responsible Party: Gordana Gedin, Head Principal, Scandinavian College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/1965-31/4
Record Dates: First submitted 2010-04-09; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-04

CONDITIONS: Other Biomechanical Lesions; Talo-crural Joint Dysfunction
Keywords: Ankle joint; Talo-crural joint; Vertical jump; Chiropractic manipulation (HVLA); ROM; Proprioception; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Single high-velocity, low-amplitude (HVLA) thrust manipulation towards Tibia, not affecting the dysfunctional talo-crural joint
  Interventions: Other: Chiropractic (HVLA) manipulation
- Treatment (Experimental): Single high-velocity, low-amplitude (HVLA long axis) thrust manipulation on dysfunctional talo-crural joint
  Interventions: Other: Chiropractic (HVLA) manipulation

INTERVENTIONS:
Other: Chiropractic (HVLA) manipulation — Single high-velocity, low-amplitude (HVLA long axis) thrust manipulation to the talo-crural joint, once a week during a three week period

SUMMARY:
The purpose of this trial was to explore the effects of chiropractic manipulation in patients with talo-crural joint dysfunction.

DETAILED DESCRIPTION:
Ankle sprains is one of the most common problems in clinical practice, mostly due to loss of mobility. Factors affecting the mobility of the joints may be due to muscle tension, ligamentous or anatomical anomalies.

Research over the last years have reported a scarce of trials investigating chiropractic treatment of the ankle joint. Previous studies have focused on investigating ROM and proprioception. This study aimed to determine whether a single high-velocity, low-amplitude (HVLA) thrust manipulation to the talo-crural joint altered ankle function in subjects with dysfunction of the talo-crural joint.

ELIGIBILITY:
Inclusion Criteria:

* First league handball player
* Talo-crural joint dysfunction
* Age >16 yrs

Exclusion Criteria:

* Patients with a history of recent trauma or previous operations with remaining fixation material in the foot or ankle

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Counter movement jump; IVAR test system | Day 1
  First assessment: One leg single jump before and after treatment (active or placebo)

SECONDARY OUTCOMES:
Counter movement jump; IVAR test system | Week one
  Second assessment: Active or placebo treatment if needed
Counter movement jump; IVAR test system | Week two
  Third assessment: One leg single jump before and after treatment (active or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Håkan A Westerblad, MD, PhD, Study Director — Karolinska Institutet
Locations (1):
- Scandinavian College of Chiropractic, Solna, Stockholm County, Sweden